CLINICAL TRIAL: NCT00219388
Title: Efficacy and Safety of Short-term Intravenous Treatment With Simdax® Versus Dobutrex® in Decompensated Heart Failure Patients Treated With Beta-receptor Blocking Agents.
Brief Title: Efficacy and Safety of Treatment With Simdax® Versus Dobutrex® in Decompensated Heart Failure Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3001075; Sponsor: Orion Pharma
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2005-09

CONDITIONS: Heart Failure
Keywords: Safety; Efficacy; Levosimendan; Dobutamine; Intravenous; Invasive hemodynamics; Decompensated Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Simendan

INTERVENTIONS:
Drug: Levosimendan

SUMMARY:
The purpose of this study is to compare the effects of levosimendan with dobutamine on heart function in patients suffering of severe chronic heart failure.

DETAILED DESCRIPTION:
Patients with decompensate heart failure (NYHA III-IV) and in need of intravenous inotrop support and who fulfil all inclusion and no exclusion criteria will be randomised into the study in proportion 1:1. Although stratification will be done so patients treated with beta-receptor blocker carvedilol will be divided the same between the study groups.

All patients will receive infusions in parallell, one of the groups will receive active product (levosimendan or dobutamine) and the other will receive placebo (double-dummy technique).

Catheterisation for measurement of hemodynamic parameters will be performed according to routine methods at the clinic. The measurements of the hemodynamic variables will start 30 minutes before start of study drug infusion and will be finished 48 hours after start of infusion. The most important variables during the measurements is Cardiac Index (CI)and Pulmonary Capillary Wedge Pressure (PCWP).

Parallel registration will be done on ECG, blood pressure, blood frequency, central venous pressure, and lung artery pressure. Heart failure and other clinical symptoms will be registered continuously during 48 hours. Blood samples will be taken intermittent to record the blood values. Cogent rules for decreasing/increasing of the dose can be found in the study protocol, likewise rules for interruption or stoop for infusion.

Registration of side-effects will be done continuously. The recommendation for treatment for known side effects could be found in the protocol (section 5.3.4) and the protocol should be available during the study procedure.

One month after the study the patients will be followed up with a very careful examination and also of the amount of visits and reason for visits to hospital during the past 30-35 days.

ELIGIBILITY:
Main Inclusion Criteria:

* Decompensated chronic heart failure of ischemic or non-ischemic origin, in NYHA class III to IV, despite optimised conventional treatment and who may benefit from intravenous positive inotropic agents as per the investigator's judgment.
* Ongoing treatment with a beta-receptor blocking agent in a stable regimen for at least 3 months and at an optimal dose as per the investigator's judgment.
* Left ventricular (LV) ejection fraction (EF) less than or similar to 35%.
* CI < 2.5 l/min/m2.
* Mean PCWP >15 mmHg.

Main Exclusion Criteria:

* Significant mechanical obstruction affecting ventricular filling and/or outflow.
* Systolic blood pressure 85 mmHg or less at screening and/or baseline.
* Heart rate 130 bpm or greater, persistent for at least 5 minutes at screening and/or baseline.
* Severe angina pectoris during the 6 hours before screening and/or baseline.
* Deterioration of chronic heart failure due to an acute myocardial infarction within 5 days before screening measurements.
* Administration of Simdax within 1 month before baseline.
* A history of Torsades de Pointes.
* Evidence of severe renal insufficiency (serum creatinine > 450 μmol/l or on dialysis) at screening.
* Significant hepatic impairment or elevation of liver enzymes to 5 times the upper limit of normal range of the analysing laboratory at screening.
* Acute bleeding or severe anaemia.
* Heart surgery within 3 months before baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-11; Study Completion 2005-04

PRIMARY OUTCOMES:
Compare the hemodynamic parameters Cardiac Index (CI) and Pulmonary Capillary Wedge Pressure (PCWP) from baseline to 24 hours, between the two groups.

SECONDARY OUTCOMES:
Compare the efficacy and safety between the treatment groups, with regard to:
• Changes in hemodynamic parameters from baseline to 24 and 48 hours.
• Change in study subject's and investigator's assessment of symptoms of heart failure at 48 hours and 1-month follow-up.
• Change in New York Heart Association (NYHA) classat 48 hours and 1-month follow-up.
• Ability to continue treatment with β-receptor blocking agents.
• Days alive and out of hospital during the 1-month follow-up period.
• Change in B-type Natriuretic Polypeptide (BNP)at 24 and 48 hours and 1-month follow-up.
• Proportion of treatment discontinuations and/or need for rescue therapy due to lack of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Claes-Håkan Bergh, Assoc Prof, Principal Investigator — Institution of Cardiology, Sahlgrenska University Hospital, Sweden
Locations (1):
- Cardiology Department, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Follath F, Cleland JG, Just H, Papp JG, Scholz H, Peuhkurinen K, Harjola VP, Mitrovic V, Abdalla M, Sandell EP, Lehtonen L; Steering Committee and Investigators of the Levosimendan Infusion versus Dobutamine (LIDO) Study. Efficacy and safety of intravenous levosimendan compared with dobutamine in severe low-output heart failure (the LIDO study): a randomised double-blind trial. Lancet. 2002 Jul 20;360(9328):196-202. doi: 10.1016/s0140-6736(02)09455-2. PMID 12133653